CLINICAL TRIAL: NCT03235089
Title: A 6-Hour Clinical Evaluation of New Daily-Wear Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV-17-46
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This will be a non-dispensing, double-masked, contralateral study comparing test contact lens against a nelfilcon A control lens. Subjects will be randomized to wear the test lens in one eye and the control lens in the other. It is anticipated that this study will involve up to 2 scheduled visits, at Baseline (BL) and 6 hours.
Who Masked: Participant, Investigator
Masking Description: Both subject and investigator will be masked to lens type for each eye. A different investigator will select the study lenses for insertion by the subject, from those performing the assessments in order to maintain masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test lens (Active Comparator): Each subjects will wear a test lens in one eye and the control lens in the other as an unmatched pair, per predetermined randomization schedule (to determine which eye receives test/control lens).
  Interventions: Device: Test Lens; Device: Control Lens
- nelfilcon A lens (control) (Active Comparator): Each subjects will wear a test lens in one eye and the control lens in the other as an unmatched pair, per predetermined randomization schedule (to determine which eye receives test/control lens).
  Interventions: Device: Test Lens; Device: Control Lens

INTERVENTIONS:
Device: Test Lens — Daily disposable contact lens
Device: Control Lens — Focus Dailies All Day Comfort contact lens (nelfilcon A)

SUMMARY:
The purpose of this study is to validate the clinical performance of a new contact lens design when worn over a period of 6 hours compared to nelfilcon A (control).

DETAILED DESCRIPTION:
The purpose of this study is to validate the clinical performance of a new contact lens design when worn over a period of 6 hours compared to nelfilcon A (control). The primary outcomes of interest are lens fit and lens fit preference.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and has full legal capacity to volunteer
* Has read, fully understood and signed the information consent letter
* Currently wears or has previously worn soft contact lenses
* Has spectacle cylinder ≤1.00D in both eyes.
* Has spherical contact lens power requirement between -1.00D and -6.00D in both eyes.
* Has manifest refraction visual acuities (VA) equal to or better than logMAR equivalent of 20/25 in each eye.
* Has clear corneas and no active ocular disease
* Is willing and able to follow product usage instructions and maintain the visit schedule.

Exclusion Criteria:

* Has never worn contact lenses before
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable
* Has any known active ocular disease and/or infection
* Has a monovision correction
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses
* Is aphakic
* Has undergone corneal refractive surgery
* Is pregnant or lactating, determined by self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Test Lens: Each subjects will wear a test lens in one eye and the control lens in the other as an unmatched pair, per predetermined randomization schedule.
  Test Lens: Daily disposable contact lens
- Nelfilcon A Lens (Control): Each subjects will wear a test lens in one eye and the control lens in the other as an unmatched pair, per predetermined randomization schedule.
  Control Lens: Focus Dailies All Day Comfort contact lens (nelfilcon A)
Period: Overall Study
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Started | 31; 31 Eyes | 31; 31 Eyes
Completed | 28; 28 Eyes | 28; 28 Eyes
Not Completed | 3; 3 Eyes | 3; 3 Eyes
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear test lens in one eye and control lens in other eye for 6 hours.
Arm/Group | Overall Study
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Horizontal Lens Centration Assessed in Primary Gaze
Description: Horizontal Lens Centration assessed in primary gaze was measured in 0.1mm steps. (mm-nasal decentration given +ve value, temporal decentration given -ve value)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | -0.13 (0.20) | -0.04 (0.21)

2. Primary Outcome: Horizontal Lens Centration Assessed in Primary Gaze
Description: as for outcome 1
Time Frame: 6-hour
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | -0.15 (0.20) | -0.06 (0.16)

3. Primary Outcome: Vertical Lens Centration Assessed in Primary Gaze
Description: Vertical Lens Centration assessed in primary gaze was measured in 0.1mm steps. (mm-superior decentration given +ve value, inferior decentration given -ve value)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 0.17 (0.25) | 0.06 (0.20)

4. Primary Outcome: Vertical Lens Centration Assessed in Primary Gaze
Description: as for outcome 3
Time Frame: 6-hours
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 0.10 (0.22) | -0.03 (0.25)

5. Primary Outcome: Lens Tightness Assessed by Push-up Test
Description: Lens Tightness was assessed by Push-up test 1% steps: (0%=Falls from cornea without lid support, 50%=Optimum, 100%=No movement)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
units on a scale | 38 (7) | 41 (6)

6. Primary Outcome: Lens Tightness Assessed by Push-up Test
Description: as for outcome 5
Time Frame: 6-hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
units on a scale | 41 (8) | 49 (6)

7. Primary Outcome: Primary Gaze Lag Assessed Observing Lens Movement in Graticule
Description: Primary gaze lag was assessed observing lens movement in graticule (0.1mm steps)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 0.16 (0.06) | 0.13 (0.05)

8. Primary Outcome: Primary Gaze Lag Assessed Observing Lens Movement in Graticule
Description: Primary gaze lag was assessed observing lens movement in graticule (0.1mm steps)
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 0.18 (0.08) | 0.12 (0.04)

9. Primary Outcome: Horizontal Lens Lag Assessed Observing Lens Movement in Graticule
Description: Horizontal lens lag was assessed observing lens movement in graticule (0.1mm steps)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 3.1 (0.3) | 2.7 (0.3)

10. Primary Outcome: Horizontal Lens Lag Assessed Observing Lens Movement in Graticule
Description: Horizontal lens lag was assessed observing lens movement in graticule (0.1mm steps)
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 3.0 (0.3) | 2.7 (0.4)

11. Primary Outcome: Overall Lens Fit Acceptance
Description: Overall lens fit acceptance based on lens fit alone (scale 0-4 in 0.25 steps: 0=can't be worn, 1=Poor, 2=Fair, 3=Good, 4=Optimum)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Nelfilcon A Lens ( Control): Each subjects will wear a test lens in one eye and the control lens in the other as an unmatched pair, per predetermined randomization schedule.
  Control Lens: Focus Dailies All Day Comfort contact lens (nelfilcon A)
Arm/Group | Test Lens | Nelfilcon A Lens ( Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
units on a scale | 2.7 (0.6) | 3.1 (0.4)

12. Primary Outcome: Overall Lens Fit Acceptance
Description: as for outcome 11
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
units on a scale | 2.7 (0.5) | 3.0 (0.5)

13. Primary Outcome: Up Gaze Lag Assessed Observing Lens Movement in Graticule
Description: Up gaze lag was assessed observing lens movement in graticule (0.1mm steps) (The amount of lens drop in mm that occurs when the eye moves from primary gaze to up gaze).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 0.41 (0.18) | 0.38 (0.16)

14. Primary Outcome: Up Gaze Lag Assessed Observing Lens Movement in Graticule
Description: as for outcome 13
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 0.34 (0.11) | 0.35 (0.14)

15. Primary Outcome: Post-blink Movement Assessed by Amount of Lens Movement Immediately After the Blink
Description: Post-blink Movement was assessed by amount of movement (to the nearest 0.1mm) immediately after the blink
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 0.44 (0.14) | 0.31 (0.11)

16. Primary Outcome: Post-blink Movement Assessed by Amount of Lens Movement Immediately After the Blink
Description: Post-blink Movement was assessed by amount of movement (to the nearest 0.1mm) immediately after the blink
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 28 | 28
Number analyzed (Eyes) | 28 | 28
millimeters | 0.43 (0.17) | 0.29 (0.11)

ADVERSE EVENTS:
Time Frame: From dispense up to 6 hours on each type of study lenses
Arm/Group | Test Lens | Nelfilcon A Lens ( Control)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT03235089/Prot_SAP_000.pdf